CLINICAL TRIAL: NCT06702839
Title: Investigation of the Effects of BETY on Biopsychosocial Status, Functionality, Mood and Quality of Life of Individuals Diagnosed With Rheumatism and Related to Chronic Pain: A Retrospective Controlled Study
Brief Title: Effect of BETY on Biopsychosocial States Associated With Chronic Pain in Rheumatic Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sevim Öksüz, Asst. Prof. Dr., Eastern Mediterranean University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBA 23/196
Record Dates: First submitted 2024-11-22; First posted 2024-11-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Rheumatic Diseases
Keywords: biopsychosocial; holistic; exercise; functioning; sleep; chronic pain
MeSH Terms: conditions — Rheumatic Diseases; Motor Activity; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Exercise Therapy Approach (Bilişsel Egzersiz Terapi Yaklaşımı-BETY) (Experimental): 3 days a week for 3 months
  Interventions: Other: BETY (Cognitive Exercise Therapy Approach )
- Home exercise program (Active Comparator): For 3 months
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: BETY (Cognitive Exercise Therapy Approach ) — Individuals with rheumatism were included in BETY sessions after the first session, which included functional gain with function-focused trunk stabilization exercises for their complaints and chronic pain management training based on neuroscience. BETY sessions included function-focused trunk stabilization exercises, chronic pain management, mood information management (dance therapy - authentic movement) as innovative. Individuals were included in a separate session of sexual information management and sleep education.
  3 days a week for 3 months
  Arms: Cognitive Exercise Therapy Approach (Bilişsel Egzersiz Terapi Yaklaşımı-BETY)
Other: Home exercise program — Exercises have been shown and a brochure has been given The individuals in this group were mostly individuals from out of town who were given home exercise recommendations directed by a rheumatologist.
  Arms: Home exercise program

SUMMARY:
No study has been found in the literature investigating the effectiveness of an innovative exercise approach defined on a biopsychosocial basis and having its own original scale on individuals with rheumatism over the years. The aim of this retrospective study was to determine the effects of the Cognitive Exercise Therapy Approach on the biopsychosocial conditions related to chronic pain; functionality, mood and quality of life of individuals with rheumatism diagnosis and to examine the effectiveness of BETY as a routine exercise approach by presenting the results compared with the control group.

DETAILED DESCRIPTION:
Cognitive Exercise Therapy Approach (BETY) is an innovative exercise approach developed through the participation of rheumatic individuals in exercise sessions for many years. The main purpose of BETY is to transfer the patient's negative cognitions about their disease to a positive cognition level through functional gains through exercise. Thus, cognitive restructuring will be achieved.

In order to correctly organize the optimum treatment, rheumatic patients need to be evaluated biopsychosocially. Individual-centered scales that evaluate the disease process are currently considered at least as much as objective tests in determining treatment effectiveness and are increasingly used in clinical practice. Due to the multidimensional structure of chronic diseases, there is a need for measurement tools that evaluate individuals in a biopsychosocial context. BETY-Biopsychosocial Scale (BETY-BQ) was developed for this purpose with the feedback of the recovery characteristics of rheumatic individuals who participated in BETY sessions over the years.

ELIGIBILITY:
Inclusion Criteria:

- Patients who were diagnosed as Ankylosing spondylitis (1984 modified New York criteria, RA (2010 ACR/EULAR criteria), PsA (2006 CASPAR criteria), SLE (2012 Systemic Lupus International Collaborating Clinics criteria), SSc (2013 ACR/EULAR criteria), pSS (American-European Consensus Group criteria), OA (1986 ACR criteria) and FMS (2016 ACR criteria)

Exclusion Criteria:

* Patients who had severe cognitive problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire (BETY-BQ): | 3 months
  it is a 30-item Likert-type scale developed through repeated statistics of feedback from rheumatic individuals who have participated in exercise sessions for many years, expressing the healing characteristics. It evaluates the individual from a biopsychosocial perspective with the subheadings of pain, functionality-fatigue, mood, sociability, sexuality and sleep. It is scored between 0 and 120. BETY-BQ evaluates the individual from a holistic perspective with six subheadings: pain (5 items), functionality (9 items), mood (10 items), sociability (3 items), sexuality (2 items) and sleep (1 item). A high score indicates a low biopsychosocial status.

SECONDARY OUTCOMES:
Health Assessment Questionnaire (HAQ) | 3 months
  It is a scale developed to question functional inadequacy in daily living activities. The scale questions a total of 8 activities, including dressing, sitting up, eating, walking, hygiene, reaching out, grasping and daily tasks, and consists of 20 questions. Each question is scored between 0 and 3. High scores indicate a decrease in the individual's functionality.
Hospital Anxiety Depression Scale (HADS) | 3 months
  It is a scale consisting of 14 questions (7 questions about depression, 7 questions about anxiety) that the individual is asked to answer by thinking about the last few days, and is scored between 0 and 3. The cut-off values of the scale are 10 for the anxiety subscale and 7 for the depression subscale. High total scores indicate high levels of anxiety or depression
Short Form - 36 (SF-36) | 3 months
  SF-36, which is widely used in assessing quality of life, is a scale consisting of 8 sub-parameters: physical function (FF), social function (SF), role limitations due to physical problems, role limitations due to emotional problems, pain, energy level-vitality, mental health and general health perception. Each sub-parameter is scored between 0 and 100. High scores indicate good health status (35).

CONTACTS AND LOCATIONS:
Overall Officials: Aykut Ozçadırcı, Principal Investigator — Hacettepe University; Nur Banu Karaca, MSc. PT., Principal Investigator — Hacettepe University; Orkun Tüfekçi, MSc. PT., Principal Investigator — Hacettepe University; Aysima Barlak, Principal Investigator — Hacettepe University; Ali Akdoğan, Prof. Dr., Study Director — Hacettepe University; Sedat Kiraz, Prof. Dr., Study Director — Hacettepe University; Edibe Unal, Prof. Dr., Study Chair — Hacettepe University; Sevim Oksüz, PhD. PT., Principal Investigator — Eastern Mediterranean University; Şule Apraş Bilgen, Prof. Dr., Study Director — Hacettepe University; Robert D. Gerwin, MD., Study Director — Johns Hopkins University; Rinnie Geenen, Prof. Dr., Study Director — Utrecht University
Locations (1):
- Hacettepe University, Ankara, Samanpazar, Turkey (Türkiye)